CLINICAL TRIAL: NCT04885101
Title: Comparison of Conservative Treatment Options in the Management of Erectile Dysfunction: Randomized Controlled Clinical Trial
Brief Title: Comparison of Conservative Treatment Options in the Management of Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Collaborators: Indústria Brasileira Equipamentos Médicos - IBRAMED (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAP DE
Record Dates: First submitted 2020-11-24; First posted 2021-05-13 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Erectile Dysfunction
Keywords: Extracorporeal Shockwave Therapy; Radiofrequency Therapy
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: The study will be conducted men diagnosed with Erectile Dysfunction alocated in three groups: Non-Ablative Radiofrequency Therapy (NARFT), Low Intensity Shockwave Therapy (LISWT) or Sham.
Who Masked: Investigator
Masking Description: The investigator won't be aware where participants will be allocated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LISWT Group (Experimental): Participants who will submitted to active procedure with Low Intensuty Shockwave Therapy.
  Interventions: Procedure: LISWT Group
- NARFT Group (Experimental): Participants who will submitted to active procedure with Non-Ablative Radiofrequency Therapy
  Interventions: Procedure: NARFT Group
- Sham Group (Sham Comparator): Participants who submitted to sham procedure with vaccum therapy.
  Interventions: Procedure: Sham Group

INTERVENTIONS:
Procedure: LISWT Group — The treatment consists of a weekly session and 4,000 pulses will be emitted each of the eight sessions totaling 32,000 pulses with a frequency of 18Hz and 100mJ of energy.
  Arms: LISWT Group
Procedure: NARFT Group — The device used will be with an intensity of 350 Wpp; 75% pulsed operation mode; frequency of 640 kHz, 1200 kHz and 2400 kHz. Eight radio frequency sessions will be held with an interval of seven days between them.
  Arms: NARFT Group
Procedure: Sham Group — In the RNA group, radiofrequency will be applied, the device used will be the Nèartek Esthetic Ibramed - Tecarterapia e Radiofrequency Apparatus, with an intensity of 350 Wpp; 75% pulsed operation mode; frequency of 640 kHz, 1200 kHz and 2400 kHz. The radiofrequency will be applied with the patient in the supine position on both sides of the penis with an opposite dispersion plate against the radiofrequency emitter. To perform the procedure, the therapist will use a glove. Eight radio frequency sessions will be held with an interval of seven days between them.
  Arms: Sham Group

SUMMARY:
This is a randomized clinical trial study with the formation of three groups. After signing the informed consent form, in two copies of equal content, the patient will be evaluated by an experienced physiotherapist and will answer a questionnaire of socio-demographic data and basic anamnesis.

Then, in a private and individualized room, participants will be guided by researchers trained to complete the self-administered questionnaires: International Erectile Function Index (IIFE), Erection Quality Questionnaire (EQQ), SF-36 and Hospital Anxiety Scale and Depression (EHAD). After applying the questionnaires, a physical evaluation by an experienced physiotherapist will be performed.

To induce erection of the penis an injection of a vasoactive agent (prostaglandin E1, alprostadil) will be administered in the corpora cavernosa. Then the length of the penis (swollen, elongated and flaccid) and penile circumference will be measured. Soon after, Dynamic Doppler Ultrasonography with Penis Doppler (UDDP) will be performed. The parameters that will be used in the UDDP to provide a general vascular diagnosis include Peak Systolic Speed (VSP), Final Diastolic Speed (VDF) and Resistive Index (IR).

In the case of a controlled and randomized clinical trial, the patient may be randomly allocated to one of three groups: the Non-Ablative Radiofrequency group (NARFT); the Low Intensity Shockwave Therapy Group (LISWT) and; the Sham Group that will perform the Vacuum Therapy (SHAM). In the NARFT group, the radio frequency will be applied, the device used will be the HERTIX Radiofrequency. The shock wave therapy application protocol in the LISWT group will use the THORK Shock Wave. While in the SHAM group, the vacuum therapy will be used, the research subjects will use the automatic version with simple on / off and release valve commands.

As in the other groups, participants in the Sham group will have a session every seven days for eight weeks. The entire evaluation protocol will be applied before (pre-test) and after treatment (post-test).

ELIGIBILITY:
Inclusion Criteria:

* 30-80 years.
* Men with a report of complaints of erectile dysfunction.

Exclusion Criteria:

* History of neurological disease.
* History of diabetes mellitus.
* History of Peyronie's disease.
* History of psychiatric illness.
* History of prostatectomy.
* Patients with anatomical malformations in the genital region.
* Penile prosthesis users.

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in peak systolic velocity | Change from baseline peak systolic velocity immediately after intervention.
  Performed by means of ultrasonography with doppler of the penis through the induction of the erection, being considered arterial insufficiency the value below 25 cm / s
Change in end diastolic velocity | Change from baseline end diastolic velocity immediately after intervention.
  Performed by means of ultrasonography with doppler of the penis through the induction of the erection, being considered venous occlusive disease the value above 5 cm / s
Change in cavernous artery diameter | Change from baseline cavernous artery diameter immediately after intervention.
  Performed by means of ultrasonography with doppler of the penis through the induction of the erection.

SECONDARY OUTCOMES:
Change in International Index of Erectile Function | Change from baseline International Index of Erectile Function immediately after intervention.
  It is a questionnaire with 5 questions about penile erection that can vary from 5 to 25 points. Higher scores indicate better clinical condition.
Change in Questionnaire of Erectile Quality | Change from baseline Questionannaire of Erectile Quality immediately after intervention.
  It is a questionnaire with 6 questions about the quality of erection based on the Likert scale. That is, it does not offer number values.
Change in measurement of penis length and diameter. | Change from baseline measurement of penis lenght and diameter immediately after intervention.
  These measurements are made with a paper ruler with the penis flaccid and after ten minutes of induction for erection.

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia V Lordêlo, PhD, Study Chair — Centro de Atenção Pélvica - CAAP
Locations (1):
- Centro de Atenção ao Assoalho Pelvico, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Background] NIH Consensus Conference. Impotence. NIH Consensus Development Panel on Impotence. JAMA. 1993 Jul 7;270(1):83-90. No abstract available. PMID 8510302
- [Background] McMahon CG, Abdo C, Incrocci L, Perelman M, Rowland D, Waldinger M, Xin ZC. Disorders of orgasm and ejaculation in men. J Sex Med. 2004 Jul;1(1):58-65. doi: 10.1111/j.1743-6109.2004.10109.x. PMID 16422984
- [Background] Mobley DF, Khera M, Baum N. Recent advances in the treatment of erectile dysfunction. Postgrad Med J. 2017 Nov;93(1105):679-685. doi: 10.1136/postgradmedj-2016-134073. Epub 2017 Jul 27. PMID 28751439
- [Background] Feldman HA, Goldstein I, Hatzichristou DG, Krane RJ, McKinlay JB. Impotence and its medical and psychosocial correlates: results of the Massachusetts Male Aging Study. J Urol. 1994 Jan;151(1):54-61. doi: 10.1016/s0022-5347(17)34871-1. PMID 8254833
- [Background] Stein RA. Endothelial dysfunction, erectile dysfunction, and coronary heart disease: the pathophysiologic and clinical linkage. Rev Urol. 2003;5 Suppl 7(Suppl 7):S21-7. PMID 16985979
- [Background] Feldman HA, Johannes CB, Derby CA, Kleinman KP, Mohr BA, Araujo AB, McKinlay JB. Erectile dysfunction and coronary risk factors: prospective results from the Massachusetts male aging study. Prev Med. 2000 Apr;30(4):328-38. doi: 10.1006/pmed.2000.0643. PMID 10731462
- [Background] Mobley D, Baum N. Smoking: Its Impact on Urologic Health. Rev Urol. 2015;17(4):220-5. PMID 26839519
- [Background] Wespes E, Amar E, Hatzichristou D, Hatzimouratidis K, Montorsi F, Pryor J, Vardi Y; EAU. EAU Guidelines on erectile dysfunction: an update. Eur Urol. 2006 May;49(5):806-15. doi: 10.1016/j.eururo.2006.01.028. Epub 2006 Feb 9. PMID 16530932
- [Background] Porst H, Burnett A, Brock G, Ghanem H, Giuliano F, Glina S, Hellstrom W, Martin-Morales A, Salonia A, Sharlip I; ISSM Standards Committee for Sexual Medicine. SOP conservative (medical and mechanical) treatment of erectile dysfunction. J Sex Med. 2013 Jan;10(1):130-71. doi: 10.1111/jsm.12023. PMID 23343170
- [Background] Chaussy C, Brendel W, Schmiedt E. Extracorporeally induced destruction of kidney stones by shock waves. Lancet. 1980 Dec 13;2(8207):1265-8. doi: 10.1016/s0140-6736(80)92335-1. PMID 6108446
- [Background] Chung E, Wang J. A state-of-art review of low intensity extracorporeal shock wave therapy and lithotripter machines for the treatment of erectile dysfunction. Expert Rev Med Devices. 2017 Dec;14(12):929-934. doi: 10.1080/17434440.2017.1403897. Epub 2017 Nov 29. PMID 29119841